CLINICAL TRIAL: NCT04666051
Title: Is There a Role for Fibrin Glue (Sealant) in Seroma Reduction After Inguinal Lymphadenectomy?
Brief Title: Fibrin Glue in Inguinal Lymphadenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, M. Ashraf Balbaa, Associate Professor of Surgery, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4/2015/SURG
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Seroma
Keywords: Fibrin glue; Seroma; Inguinal lymphadenectomy; Wound complication
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Fibrin glue (Experimental): A fibrin glue was applied to the lymphadenectomy bed before wound closure and insertion of a drain.
  Interventions: Biological: Application of fibrin glue sealant
- Control (No Intervention): Lymphadenctomy wound was closed after insertion of a drain,

INTERVENTIONS:
Biological: Application of fibrin glue sealant
  Arms: Fibrin glue

SUMMARY:
Seroma is one of the most common encountered morbidities after inguinal lymph node dissection (ILND). It can cause not only much nuisance to both patients and doctors but also its presence can lead to many complications. This study aimed at evaluation of the role and effect of using fibrin glue on seroma reduction in patients undergoing ILND. Thirty-two patient have undergone ILND for various causes. The patients were randomized into two groups; 16 ILND in each. In one group, fibrin glue sealant was applied with a dose of 2ml per 100 cm2 surface area then drain placement was performed. Whereas, in the control group, only drain placement was used. Preoperative, operative and postoperative data were recorded and analyzed.

DETAILED DESCRIPTION:
Seroma is one of the most frequent complications occurring after ILND as it affects nearly one third of these cases. During the past decades, many actions have been tried in the perioperative care to decrease the incidence of these complications, as employing well vascularized bulky flaps to obliterate the dead space and to protect vessels, great saphenous vein sparing, strict bed rest and fibrin sealant application. Realizing the underlying pathology for seroma formation is the key point in its prevention. Thirty-nine patients scheduled to perform Inguinal lymphadenectomy for various causes have been checked for eligibility to be enrolled in this prospective, randomized study. Thirty-two patients have met the inclusion criteria. Inguinal lymphadenectomy has been performed including scarifying saphenous vein. Sartorius muscle transposition flap was routinely performed for protection of femoral vessels, then an 18 French conventional non-suction tube drain was inserted in all patients. All the previous steps were similar in both groups. At this stage, the wound was closed for the control group, while fibrin glue was prepared to be applied to the fibrin glue group in a dose of 2mL for 100 cm2 surface area. Postoperatively, the daily collected drain fluid was measured till the drain was removed when the daily drainage was less than 30 ml. Then the patients were planned to be followed up postoperatively for at least 4 weeks, to detect the possible clinically encountered complications as seroma, wound infection, or skin flap necrosis.

Patients' demographic data and preexisting co-morbidities were recorded. Operative and pathological data regarding defect size, blood transfusion, primary tumor pathology, and number and status of retrieved lymph nodes were collected. The occurrence of post-operative seroma was the primary outcome. Other non serious adverse effect as hematoma, infection, or skin flap necrosis were recorded and compared between the two groups.

The normality of distribution of variables was verified by Kolmogorov- Smirnov test. Chi-square test (Fisher or Monte Carlo) was used for comparisons between groups for categorical variables. Student t-test was used to compare two groups for normally distributed quantitative variables. For not normally distributed quantitative variables, Mann Whitney test was used to compare between two groups. P value was set to be significant if <0.05.

ELIGIBILITY:
Inclusion Criteria:

• Patients scheduled to perform ILND for various causes

Exclusion Criteria:

* BMI more than 35,
* Uncompensated diabetes
* Advanced liver disease
* Previous history of surgery and/or irradiation to the inguinal region
* Preoperative chemotherapy
* Significant coagulation disorders
* Platelet counts <100,000/mL.
* Use of systemic steroids or anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Ashraf Balbaa, M.D., Study Director — Menoufia University

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be available to be shared on request after study publication for 6 months.
Supporting Information: Study Protocol
Time Frame: Six months from the time of study publication
Access Criteria: Contacting the corresponding author

REFERENCES:
- [Background] Buda A, Fruscio R, Pirovano C, Signorelli M, Betti M, Milani R. The use of TachoSil for the prevention of postoperative complications after groin dissection in cases of gynecologic malignancy. Int J Gynaecol Obstet. 2012 Jun;117(3):217-9. doi: 10.1016/j.ijgo.2011.12.021. Epub 2012 Mar 15. PMID 22424660

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibrin Glue: A fibrin glue was applied to the lymphadenectomy bed before wound closure and insertion of a drain.
  Application of fibrin glue sealant
Period: Overall Study
Arm/Group | Fibrin Glue | Control
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Glue | Control | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.40 (8.16) | 55.94 (8.1) | 56.19 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 16 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 16 | 16 | 32
Inguinal lymphadenectomy [Number; unit: participants] | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroma Formation
Description: Collection of serous fluid under the wound flaps. According to the Common Terminology Criteria for Adverse Events (CTCAE) 4.0, Grade 2 and Grade 3 were considered.
  Grade 2 indicates it is symptomatic; simple aspiration indicated. Grade 3 indicates it is symptomatic, elective radiologic or operative intervention indicated
Time Frame: 4 weeks postpertively
Population: Serum formation has been looked for
Measure: Number; unit: participants
Arm/Group | Fibrin Glue | Control
Number analyzed (Participants) | 16 | 16
participants | 2 | 8
Statistical Analysis 1: Comparison: Fibrin Glue vs Control; Test type: Superiority — Data from both groups has been collected compared to verify significant statistical difference; p = 0.022, Chi-squared

ADVERSE EVENTS:
Time Frame: The follow up period ranged from 4 to 8 weeks with a median of 4 weeks.
Description: Hematoma, infection and partial superficial skin edge necrosis have been recorded as adverse effects that are categorized as "Other" adverse effects as per clinical trails.gov definitions,
Arm/Group | Fibrin Glue | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrin Glue (N=16) | Control (N=16)
Hematoma (Surgical and medical procedures) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 4 (4)
Partial superficial skin edge necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04666051/Prot_SAP_000.pdf